CLINICAL TRIAL: NCT01273116
Title: Towards an In Hospital CARE AND WELFARE STANDARD for Frail Elderly
Brief Title: In Hospital Care and Welfare Standard
Acronym: CWSInHosp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Marcel Olde Rikkert, prof dr, Radboud University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Nr. 60-61900-98-272, NPO
Record Dates: First submitted 2010-12-28; First posted 2011-01-10 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Functional Decline and Complications of Frail Older Patients Admitted to Hospital
Keywords: frailty; integrated care; hospital; geriatrics; hospital-wide intervention
MeSH Terms: conditions — Frailty | interventions — Hospitals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CWS in Hospital (Experimental): CWS in Hospital in addition to usual care
  Interventions: Other: CWS in Hospital

INTERVENTIONS:
Other: CWS in Hospital — Every patient aged ≥70 years will be screened for frailty. (For) every frail patient:
  * will have a comprehensive (geriatric) assessment using an adapted version of the EasyCare instrument;
  * a geriatric consultation team will propose/recommend a tailored care and welfare plan, which will be updated at the moment of discharge;
  * will be discussed at least once in a multidisciplinary meeting;
  * a structured medication review will be carried out by a geriatrician;
  * is offered an activation programme by volunteers focusing on improvement of orientation, mobility, social activities or nutrition;
  * may receive a consult of a geriatrician, if judged necessary;
  * will receive extra attention on discharge arrangements.
  Hospital staff will be educated, disease-specific guidelines will be adapted to frail older patients.

SUMMARY:
The current organization of hospital care for older patients with complex healthcare needs is of insufficient quality, safety and efficiency. Frail older patients have a higher risk for development of complications and consequently a higher length of hospital stay, a higher risk of functional decline, and higher care needs after discharge. As nearly half of the patients admitted to Dutch hospitals is over 65 years, it is highly necessary to adapt the organization of hospital care to their needs. Besides having introduced the medical specialty geriatrics, hospital management has not started to provide hospital wide healthcare tailored to frail older patients. Therefore, the purpose of this study is to develop and examine the effectiveness of an intervention program for frail older patients admitted to hospital aimed at preventing functional decline and other hospital related negative outcomes.

DETAILED DESCRIPTION:
The long-term objective of this study is to examine the effectiveness and efficiency of an intervention program for frail older patients admitted to hospital. The specific aims are:

* To develop a model of integrated hospital care, according to the principle of the Chronic Care Model, focusing both on optimizing care and wellbeing. Feasibility of such a model of care was first evaluated in a pilot study.
* To conduct a before-after study to evaluate the outcomes associated with the proposed model of hospital care in frail older inpatients. Information on outcome indicators, including autonomy, quality of life, physical and cognitive functioning, and service utilization will be collected and compared before and after implementation of the proposed model of hospital care.

We expect that older patients who participate in the intervention program after one year of implementation, compared to patients who were admitted to hospital before implementation of the intervention program, will:

* have less functional decline during admission and after three months follow-up compared to two weeks before admission;
* have a lower incidence, severity and duration of delirium during admission;
* have less cognitive decline during admission;
* are more likely to be discharged directly to their own homes;
* have less weight loss between admission and discharge;
* experience less falls during admission;
* experience less readmissions within one month after discharge;
* have a shorter length of stay;
* have a significant different pattern of use of health care services after three months follow-up;
* experience more autonomy during hospital admission and better quality of life after three months follow-up.

Additionally, we expect that the knowledge and attitudes toward care for older patients among nurses and physicians will change positively during implementation of the intervention program.

ELIGIBILITY:
Inclusion Criteria:

* Frail patients aged 70 years or older, admitted to one of the participating hospital wards
* Patients aged <70 years, but living in a nursing home or diagnosed with dementia (and therefore also judged as frail)

Exclusion Criteria:

* Patients admitted <48 hours
* Palliative care is main goal of hospital admission
* Patients admitted and treated by physicians from non-participating wards and specialities
* Patients who do not speak or understand the Dutch language

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 404 (Actual)
Dates: Start 2011-01; Primary Completion 2012-07 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Patient safety | during hospital stay
  cumulative incidence in delirium, falls, functional decline (GARS), and loss of cognition (MMSE)

SECONDARY OUTCOMES:
Maintenance or improvement of functional status (patient safety) | 2 weeks before admission, discharge, 3 months after discharge
  maintenance or improvement of functional status (Groningen Activity Restriction Scale GARS)):
  * difference between 2 weeks before admission and discharge
  * difference between discharge and 3 months after discharge
  * difference between 2 weeks before admission and 3 months after discharge
Incidence delirium (patient safety) | during hospital stay
  incidence delirium (as judged by an independent physician, structured by daily application of the Confusion Assessment Method (CAM) and Delirium Observation Scale (DOS))
Autonomy of patient (quality of care) | before implementation and one year after implementation of CWS InHospital
  Consumer Quality Indicator CWS In Hospital: to address autonomy of patients, developed by own researchers
OPROCS (quality of care) | discharge and 3 months follow-up
  OPROCS = cumulative outcome measure functional ability and quality of life etc. as determined by the elderly (Minimum Data Set)
Validity of delirium diagnoses by the medical specialty involved (quality of care) | before and one year after implementation CWS InHospital
  recognition of delirium by medical staff (nurses and doctors) compared to diagnoses by independent physician using CAM and DRS-r-98
Readmissions (quality of care) | within 1 month after discharge
  readmissions within 1 month after discharge (Minimum Data Set, electronic health record)
Objective burden of care among informal caregivers (quality of care) | from admission to 3 months after discharge patient
  objective burden of care among informal caregivers (Minimum Data Set)
Cost-effectiveness | from admission to 3 months after discharge
  expressed in incremental cost-effectiveness ratio (length of stay; use of health care services (MDS), quality of life) primary outcomes as nominator, and expressed in costs per quality adjusted life years, all related to total health care costs from a societal perspective, from admission to three months following discharge

CONTACTS AND LOCATIONS:
Overall Officials: Marcel GM Olde Rikkert, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Bakker FC, Persoon A, Bredie SJH, van Haren-Willems J, Leferink VJ, Noyez L, Schoon Y, Olde Rikkert MGM. The CareWell in Hospital program to improve the quality of care for frail elderly inpatients: results of a before-after study with focus on surgical patients. Am J Surg. 2014 Nov;208(5):735-746. doi: 10.1016/j.amjsurg.2014.04.009. Epub 2014 Jun 27. PMID 25085385